CLINICAL TRIAL: NCT05673551
Title: A Randomized Clinical Trial of Smartphone Virtual Reality for Pain Management During Burn Care Transition
Brief Title: VR-PAT During Home Burn Dressings - Multisite
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Parkland Health and Hospital System (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Henry Xiang, Professor of Medicine and Center Director, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002851
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Burns; Acute Pain; Procedural Pain; Injuries; Pediatric ALL
Keywords: Virtual Reality; VR; Burns; Pain
MeSH Terms: conditions — Burns; Acute Pain; Pain, Procedural; Wounds and Injuries; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants will be using the VR-PAT during burn dressings.
  Interventions: Other: VR-PAT
- Control Group (No Intervention): Participants will not be using the VR-PAT during burn dressings (other distraction methods available in the home allowed).

INTERVENTIONS:
Other: VR-PAT — Smartphone-based Virtual Reality Pain Alleviation Tool (VR-PAT) via a lightweight, mobile VR headset
  Other Names: Virtual Reality
  Arms: Intervention Group

SUMMARY:
This study will evaluate the effectiveness of smartphone Virtual Reality Pain Alleviation Therapy (VR-PAT) as a pain distraction tool during repeated at-home burn dressing changes among 100 children (age 6-17 years) with a burn injury in comparison to 100 children with a burn injury who do not use the VR-PAT.

DETAILED DESCRIPTION:
In this two-group randomized clinical trial, participants will be randomly assigned to either the VR-PAT intervention group or control group (standard distraction techniques available in the home). Participants and caregivers in both groups will perform daily burn dressing changes (as prescribed by their physician) and afterward will answer questions about their pain and any medications used. Participants and caregivers in the intervention group will answer additional questions about their experience using the VR-PAT, ease of use, and helpfulness. Surveys will be repeated with each dressing changes for one week.

ELIGIBILITY:
Inclusion Criteria:

* Being treated for acute burn injury
* Age 6-17 years, inclusive
* Receiving their first outpatient clinic dressing change or being discharged from the ED or inpatient burn unit
* Have a dressing that requires daily changes at home for at least 7 days after their first outpatient appointment or discharge from the hospital (ED or inpatient)
* Patient and family caregivers can communicate (read and write) using English or Spanish
* Reported at least moderate or worse NRS pain score of ≥3 (NRS 0-10 with 10 being worst pain) from the most recent dressing change.

Exclusion Criteria:

* Any wounds that may interfere with study procedures
* Vision, hearing, or cognitive/motor impairments preventing valid administration of study measures
* History of motion sickness, seizure disorder, dizziness, or migraine headaches precipitated by visual auras
* Minors in foster care, prisoners, or currently pregnant
* Suspected child abuse
* Families who do not have access to a VR compatible smartphone.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported pain | Immediately following each dressing change for one week
  0-10 Numerical Rating Scale (NRS) (self-reported and caregiver-reported), 0(min)-10(max), with higher score indicating worse pain. Asked for worst pain, average pain, and time spent thinking about pain.

SECONDARY OUTCOMES:
Self-reported VR experience | Immediately following each dressing change for one week
  0-10 Numerical Rating Scale (NRS) (self-reported - VR-PAT arm only), 0(min)-10(max), with higher score meaning better outcome. Asked for degree of realism, pleasure, and satisfaction with VR.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Parkland Health & Hospital System, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu A, Armstrong M, Alexander R, Vest E, Chang J, Zhu M, Xiang H. Trends in pediatric prescription-opioid overdoses in U.S. emergency departments from 2008-2020: An epidemiologic study of pediatric opioid overdose ED visits. PLoS One. 2024 Apr 17;19(4):e0299163. doi: 10.1371/journal.pone.0299163. eCollection 2024. PMID 38630653
- [Derived] Armstrong M, Price A, Coffey R, Noffsinger D, Thakkar RK, Fabia RB, Groner JI, Mandell S, Ni A, Xiang H. Smartphone virtual reality for pain management during pediatric burn care transition: study protocol for a randomized controlled trial. Trials. 2025 May 13;26(1):157. doi: 10.1186/s13063-025-08860-4. PMID 40361220